CLINICAL TRIAL: NCT03739684
Title: A Phase 3, Multi-Center, Open-Label Study to Assess the Diagnostic Performance and Clinical Impact of 18F-DCFPyL PET/CT Imaging Results in Men With Suspected Recurrence of Prostate Cancer
Brief Title: Study of 18F-DCFPyL PET/CT Imaging in Patients With Suspected Recurrence of Prostate Cancer
Acronym: CONDOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PyL 3301
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Cancer Recurrent; Prostate Cancer Metastatic
Keywords: Positron emission tomography; biochemical recurrence; rising PSA; PET/CT; Diagnostic; Imaging; PSMA; radical prostatectomy; BCR
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL Injection (Experimental): 9 mCi (333 MBq) IV injection of 18F-DCFPyL
  Interventions: Drug: 18F-DCFPyL; Diagnostic Test: PET/CT Imaging

INTERVENTIONS:
Drug: 18F-DCFPyL — A single dose of 9 mCi (333 MBq) IV injection of 18F-DCFPyL
  Other Names: PyL
Diagnostic Test: PET/CT Imaging — PET/CT imaging will be acquired 1-2 hours post-PyL injection

SUMMARY:
This study evaluates the diagnostic performance and safety of 18F-DCFPyL (PyL) PET/CT imaging in patients with suspected recurrence of prostate cancer who have negative or equivocal findings on conventional imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male >/= 18 years of age
* Histopathologically confirmed prostate adenocarcinoma per original diagnosis, with subsequent definitive therapy
* Suspected recurrence of prostate cancer based on rising PSA after definitive therapy on the basis of:

  1. Post-radical prostatectomy: Detectable or rising PSA that is ≥ 0.2 ng/mL with a confirmatory PSA ≥ 0.2 ng/mL (American Urological Association [AUA]); or
  2. Post-radiation therapy, cryotherapy, or brachytherapy: Increase in PSA level that is elevated by ≥ 2 ng/mL above the nadir (American Society for Therapeutic Radiology and Oncology [ASTRO]-Phoenix)
* Negative or equivocal findings for prostate cancer on conventional imaging performed as part of standard of care workup within 60 days prior to Day 1
* Life expectancy ≥6 months as determined by the investigator
* Able and willing to provide informed consent and comply with protocol requirements

Exclusion Criteria:

* Subjects administered any high energy (>300 KeV) gamma-emitting radioisotope within five (5) physical half-lives prior to Day 1
* Ongoing treatment with any systemic therapy (e.g. ADT, antiandrogen, GnRH, LHRH agonist or antagonist) for prostate cancer
* Treatment with ADT in the past 3 months of Day 1
* Receipt of investigational therapy for prostate cancer within 60 days of Day 1
* Subjects with any medical condition or other circumstances that, in the opinion of the investigator, compromise the safety or compliance of the subject to produce reliable data or completing the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males subjects will be enrolled in this study.
Enrollment: 208 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D Jensen, Study Director — Progenics Pharmaceuticals, Inc.
Locations (14):
- United States (13):
  - City of Hope National Medical Center, Duarte, California
  - Tower Urology, Los Angeles, California
  - University of California San Francisco - Helen Diller Cancer Center, San Francisco, California
  - Stanford, Stanford, California
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
- Chu de Quebec - Universite Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 18F-DCFPyL Injection: Participants with suspected recurrence of prostate cancer and negative or equivocal findings per institutional standard of care conventional imaging were enrolled to receive a single dose of 9 mCi (333 MBq) 18F-DCFPyL injection followed by a single PET/CT scan acquired 1 to 2 hours post-dosing.
Period: Overall Study
Arm/Group | 18F-DCFPyL Injection
Started | 208
Completed | 195
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: Safety population; all participants who received any amount of 18F-DCFPyL
Arm/Group | 18F-DCFPyL Injection
Number analyzed (Participants) | 208
Age, Continuous [Median (Full Range); unit: years] | 68 [43 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 208
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Black or African American | 15
  White | 188
  Other, including not reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Correct Localization Rate (CLR)
Description: The Correct Localization Rate (CLR) will be defined as percentage of participants with a one-to-one correspondence between localization of at least one lesion identified on 18F-DCFPyL PET/CT imaging and the composite truth standard. Within 60 days following PyL PET/CT imaging, either biopsy/surgery, conventional imaging, or locoregional radiation therapy of the PyL-suspected lesion(s) will be performed.
Time Frame: Within 60 days following 18F-DCFPyL PET/CT imaging.
Population: Participants who received any amount of 18F-DCFPyL and had a 18F-DCFPyL PET/CT central imaging reader result.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 18F-DCFPyL Injection
Number analyzed (Participants) | 208
percentage of participants
  Central Reader 1 | 85.6 [78.8 to 92.3]
  Central Reader 2 | 87.0 [80.4 to 93.6]
  Central Reader 3 | 84.8 [77.8 to 91.9]

2. Secondary Outcome: Percentage of Participants With a Change in Intended Prostate Cancer Treatment Plans Due to 18F-DCFPyL PET/CT Imaging Results.
Description: The change in the intended prostate cancer treatment plan will be based on Medical Management Questionnaires completed prior to and after 18F-DCFPyL PET/CT imaging.
Time Frame: Pre 18F-DCFPyL PET/CT imaging and within 60 days following 18F-DCFPyL PET/CT imaging.
Population: Participants with a Medical Management Questionnaire (MMQ) completed at pre- and post- 18F-DCFPyL PET/CT imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DCFPyL Injection
Number analyzed (Participants) | 205
Participants | 131

3. Secondary Outcome: The Change From Pre- to Post- 18F-DCFPyl Dosing in Blood Pressure (Safety Outcome Measure)
Description: The recorded values and their respective changes from the pre-dose values will be summarized using descriptive statistics.
Time Frame: Measured at 2 intervals on the day of dosing; the first interval prior to receiving the 18F-DCFPyL dose and the second interval within 60 to 120 minutes after dosing.
Population: The Safety Set includes all participants who received any amount of 18F-DECPyL.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 18F-DCFPyL Injection
Number analyzed (Participants) | 208
mmHg
  Systolic Blood Pressure: Baseline (actual): number analyzed (Participants) | 207
  Systolic Blood Pressure: Baseline (actual) | 138.9 (18.61)
  Systolic Blood Pressure: Post-dosing (actual): number analyzed (Participants) | 202
  Systolic Blood Pressure: Post-dosing (actual) | 136.7 (17.15)
  Systolic Blood Pressure: Change from Baseline: number analyzed (Participants) | 202
  Systolic Blood Pressure: Change from Baseline | -2.2 (13.24)
  Diastolic Blood Pressure: Baseline (actual): number analyzed (Participants) | 207
  Diastolic Blood Pressure: Baseline (actual) | 78.5 (10.18)
  Diastolic Blood Pressure: Post-dosing (actual): number analyzed (Participants) | 202
  Diastolic Blood Pressure: Post-dosing (actual) | 77.3 (9.57)
  Diastolic Blood Pressure: Change from Baseline: number analyzed (Participants) | 202
  Diastolic Blood Pressure: Change from Baseline | -1.2 (8.20)

4. Secondary Outcome: The Change From Pre- to Post- 18F-DCFPyL Dosing in Heart Rate (Safety Outcome Measure)
Description: as for outcome 3
Time Frame: as for outcome 3
Population: The Safety Set includes all participants who received any amount of 18F-DCFPyL.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 18F-DCFPyL Injection
Number analyzed (Participants) | 208
bpm
  Heart Rate: Baseline (actual): number analyzed (Participants) | 207
  Heart Rate: Baseline (actual) | 69.3 (12.75)
  Heart Rate: Post-dosing (actual): number analyzed (Participants) | 202
  Heart Rate: Post-dosing (actual) | 65.1 (12.09)
  Heart Rate: Change from Baseline: number analyzed (Participants) | 202
  Heart Rate: Change from Baseline | -4.3 (7.93)

5. Secondary Outcome: Collection of Concomitant Medications (Safety Outcome Measure)
Description: Medications will be coded using the WHO drug dictionary. The medications are summarized by ATC level 4 category and presented as number and percentage of participants.
  Results are presented where the percentage of participants within an ATC level 4 category is >5.0.
Time Frame: From the time of 18F-DCFPyL dosing to completion of the follow-up visit at 7 (±3) days after 18F-DCFPyL dosing.
Population: The Safety Set includes all participants who received any amount of 18F-DCFPyL.
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DCFPyL Injection
Number analyzed (Participants) | 208
Participants
  HMG COA REDUCTASE INHIBITORS | 103
  PLATELET AGGREGATION INHIBITORS (EXCLUDING HEPARIN) | 63
  ACE INHIBITORS, PLAIN | 36
  VITAMIN D AND ANALOGUES | 32
  ANGIOTENSIN II ANTAGONISTS, PLAIN | 31
  BETA BLOCKING AGENTS, SELECTIVE | 31
  DIHYDROPYRIDINE DERIVATIVES | 31
  PROTEIN PUMP INHIBITORS | 29
  DRUGS USED IN ERECTILE DYSFUNCTION | 23
  MULTIVITAMINS, PLAIN | 18
  BIGUANIDES | 17
  THIAZIDES, PLAIN | 16
  OTHER ANTIDEPRESSANTS | 15
  ALPHA-ADRENORECEPTOR ANTAGONISTS | 12
  PROPIONIC ACID DERIVATIVES | 12
  THYROID HORMONES | 11
  UNSPECIFIED HERBAL AND TRADITIONAL MEDICINE | 11

6. Secondary Outcome: Collection of Medical Procedures (Safety Outcome Measure)
Description: Procedures will be coded using the same version of MedDRA as for medical history. Medical procedures will be displayed as a listing by participant.
Time Frame: From the time of 18F-DCFPyL dosing to completion of the follow-up visit at 7 (±3) days after 18F-DCFPyL dosing.
Population: The Safety Set includes all participants who received any amount of 18F-DCFPyL.
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DCFPyL Injection
Number analyzed (Participants) | 208
Participants
  Biopsy testes | 1
  Computerized tomogram | 1
  Nuclear magnetic resonance imaging | 1
  Ultrasound testes | 1
  Open reduction of fracture | 1
  Orchidectomy | 1

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected after 18F-DCFPyL administration on Day 1 post-dose through the safety visit 7 (±3) days post-dosing.
Arm/Group | 18F-DCFPyL Injection
All-Cause Mortality (participants affected / at risk) | 0/208
Serious Adverse Events (participants affected / at risk) | 1/208
Other Adverse Events (participants affected / at risk) | 7/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 18F-DCFPyL Injection (N=208)
Hypersensitivity (Immune system disorders) | 1
Headache (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 18F-DCFPyL Injection (N=208)
Headache (Nervous system disorders) | 3
Fatigue (General disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results cannot be published before the earlier of a multi-site publication; or 18 months after the end of the Study at all sites; or confirmation by Sponsor that there will be no multi-site publication. The proposed publication must be submitted to Sponsor at least 60 days prior to publication so that Sponsor can delete Sponsor Confidential Information (other than Study results) and obtain a further 60 days to file on any invention disclosed in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT03739684/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT03739684/SAP_001.pdf